# Protocol synopsis (extracted from final protocol)



Protocol KF7039-01


SUP-006530, Rev 01

| Trial code: | KF7039-01 |
|---|---|
| Title of trial: | A randomized, double-blind, placebo-controlled, Phase III trial to evaluate the efficacy and safety of intra-articular injections of RTX-GRT7039 in adult subjects with pain associated with osteoarthritis of the knee |
| Brief title: | Comparison of RTX-GRT7039 and placebo injections for pain associated with osteoarthritis of the knee. |
| Indication: | Moderate to severe pain associated with osteoarthritis of the knee |
| International<br>Coordinating<br>Investigator: <sup>a</sup> | PPD Telephone: +PPD |
| Trial site(s): | Approximately 74 sites globally |
| | Documentation of the involved trial sites will be maintained. |
| Trial sponsor: | Grünenthal GmbH, 52099 Aachen, Germany |
| Sponsor's medically qualified person <sup>a</sup> : | PPD PPD |
| Sponsor's signatory: | PPD PPD |
| Public contact point: | Email: clinical-trials@grunenthal.com PPD |

a) Contact detail changes during the course of the trial will be documented and do not require a protocol amendment.

VersionDateDMS version numberValid forOriginal:28 Oct 20211.0All countriesUniversal TrialU1111-1268-7314EudraCT number:2021-005029-26Number:

#### CONFIDENTIAL

The contents of this document may not be disclosed to any other person without written permission from the sponsor unless required by good clinical practice or applicable regulatory requirements. Any supplemental documentation for the clinical trial is also covered by this provision.

DMS version: 1.0

ID: 1423148

Protocol synopsis 

# Protocol synopsis (extracted from final protocol)


Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

#### 1 PROTOCOL SYNOPSIS

### 1.1 Trial design

This is an interventional, Phase III, double-blind, randomized, placebo-controlled, parallel-group, multi-site, clinical trial to confirm the efficacy and safety of repeated injections of RTX-GRT7039 versus placebo in subjects who have moderate to severe pain associated with osteoarthritis of the knee despite receiving continued treatment with optimal standard of care (SoC) or who are unable to receive SoC treatment due to contraindications or intolerability.

Approximately 450 subjects will be randomized to receive either RTX-GRT7039 or placebo in a 1:1 ratio. In addition to continued SoC treatment, subjects will receive 1 of the following treatments:

- RTX-GRT7039 400 ng intra-articular injections.
- Placebo to match RTX-GRT7039 intra-articular injections.

Subjects will each receive 2 injections of investigational medicinal product (IMP) during the Double-blind Treatment Period (on Day 1 and at Week 26). For the second injection, subjects will receive the same IMP that was administered at the first injection, in a double-blind manner.

### 1.1.1 Trial design chart

See Figure 1 for an illustration of the trial design.

### Grünenthal


Protocol KF7039-01

 DMS version 1.0 28 Oct 2021





 $IA = intra-articular; \ IMP = investigational \ medicinal \ product; \ V = Visit$ 

Figure 1: Trial design chart


Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

### 1.1.2 Brief description of the sequence and duration of all trial periods

This trial comprises a Screening Period, a double-blind Treatment and Follow-up Period (including a Final Visit of the Treatment and Follow-up Period at Week 52).

Each subject is expected to be in the trial for up to 56 weeks (i.e., the Screening Period of up to 30 days followed by the 52-week Treatment and Follow-up Period).

See Section 1.1.1 for a summary of the trial design as a trial design chart and Section 1.6 for a tabular schedule of events (SoE).

### 1.2 Trial objectives and endpoints/outcomes

| Objective | Endpoint/Outcome |
|---|---|
| Primary | Primary |
| Demonstrate the analgesic efficacy of intra-articular RTX-GRT7039 compared with placebo in change from baseline at Week 12. | Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score in the index knee to the score at Week 12. The WOMAC pain subscale, which consists of 5 questions, will be assessed and reported in the electronic diary (e-diary) once weekly with a 48-hour recall, using an 11-point numeric rating scale (NRS, from 0 = no pain to 10 = pain as bad as you can imagine). Timeframe for the assessment: from baseline (assessment at V2) to V5 (Week 12/Day 84). Estimand The primary comparison of interest is the difference in mean change from baseline in 48-hour WOMAC pain subscale score at Week 12 in the index knee using an 11-point (0-10) NRS between RTX-GRT7039 and placebo, in subjects who initiate treatment, as if substantial changes in background medication or addition of new analgesics were not available. |
| Key Secondary | Key Secondary |
| Demonstrate the analgesic efficacy of intra-articular RTX-GRT7039 compared with placebo in change from baseline at Week 26 and Week 52. | Change from baseline in WOMAC pain subscale score in the index knee based on the 11-point (0-10) NRS to the score at Week 26 and at Week 52. Estimands A secondary comparison of interest is the difference in mean change from baseline in 48-hour WOMAC pain subscale score at Week 26 in the index knee using an 11-point (0-10) NRS between RTX-GRT7039 and placebo, in subjects who initiate treatment, as if substantial changes in background medication or addition of new analgesics were not available. |

### 

# Protocol synopsis (extracted from final protocol)


Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

| Objective | Endpoint/Outcome |
|---|---|
| | A secondary comparison of interest is the difference in mean change from baseline in 48-hour WOMAC pain subscale score at Week 52 in the index knee using an 11-point (0-10) NRS between RTX-GRT7039 and placebo, in subjects who initiate treatment, as if substantial changes in background medication or addition of new analgesics were not available, and as if subjects have received 2 injections with a 26-week interval (i.e., did not discontinue treatment). |
| Demonstrate the efficacy of intra-articular RTX-GRT7039 on | Change from baseline in WOMAC physical function subscale score at Week 12, at Week 26, and at Week 52. |
| function compared with placebo in change from baseline at Week 12, at Week 26, and at Week 52. | Estimand A secondary comparison of interest is the difference in mean change from baseline in 48-hour WOMAC physical function subscale score at Week 12 and at Week 26 in the index knee using an 11-point (0-10) NRS between RTX-GRT7039 and placebo, in subjects who initiate treatment, as if substantial changes in background medication or addition of new analgesics were not available. A secondary comparison of interest is the difference in mean change from baseline in 48-hour WOMAC physical function subscale score at Week 52 in the index knee using an 11-point (0-10) NRS between RTX-GRT7039 and placebo, in subjects who initiate treatment, as if substantial changes in background medication or addition of new analgesics were not available, and as if subjects have received 2 injections with a 26-week interval (i.e., did not discontinue treatment). |
| To assess the safety and tolerability of RTX-GRT7039 intra-articular injection. | Incidence of treatment-emergent adverse events (TEAEs). Incidence of TEAEs leading to discontinuation in the Treatment and Follow-up Period after the first and after the second injection, respectively. Incidence of TEAEs representing structural changes of the knee joint as visualized by the imaging methods assessed by the investigator as clinically relevant (thus constitute an adverse event [AE]) and as at least possibly related to the IMP (and not attributable to the natural progression of the disease in an individual patient). |


Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

| Objective | Endpoint/Outcome |
|---|---|
| Secondary | Secondary |
| Demonstrate the efficacy of intra-<br>articular RTX-GRT7039 compared<br>with placebo in change from baseline<br>to Week 38 in the WOMAC pain<br>subscale score and WOMAC physical<br>function subscale score. | Change from baseline in WOMAC pain subscale score and WOMAC physical function subscale score at Week 38. |
| Demonstrate the efficacy of intra-<br>articular RTX-GRT7039 compared<br>with placebo in change from baseline<br>to Week 12, to Week 26, to Week 38,<br>and to Week 52 in the WOMAC<br>stiffness subscale score, WOMAC<br>total score, and on pain when walking<br>on a flat surface (WOMAC A1). | Change from baseline in WOMAC stiffness subscale score, WOMAC total score, and pain when walking on a flat surface (WOMAC A1) at Week 12, Week 26, Week 38, and Week 52. |
| Demonstrate the efficacy of intra-<br>articular RTX-GRT7039 compared<br>with placebo in percentage of subjects<br>with ≥30%, 50%, and 70% reduction<br>in pain from baseline at Week 12, at<br>Week 26, at Week 38, and at Week 52. | Percentage of subjects with ≥30%, 50%, and 70% reduction in WOMAC pain subscale in the index knee from baseline at Week 12, from baseline at Week 26, from baseline at Week 38, and from baseline at Week 52. Percentage of subjects with ≥30%, 50%, and 70% reduction in pain when walking on a flat surface (WOMAC A1) in the index knee from baseline at Week 12, from baseline at Week 26, from baseline at Week 38, and from baseline at Week 52. |
| Demonstrate the efficacy of intra-<br>articular RTX-GRT7039 compared<br>with placebo in percentages of subjects<br>responding according to OMERACT-<br>OARSI criteria at Week 12, at<br>Week 26, at Week 38, and at Week 52. | Percent of responders according to OMERACT-OARSI criteria at Week 12, Week 26, Week 38, and Week 52. |
| Demonstrate the efficacy of intra-<br>articular RTX-GRT7039 compared<br>with placebo in patient global<br>impression of change (PGIC). | PGIC at Week 12, Week 26, Week 38, and Week 52. |
| Demonstrate the quality of life after treatment with RTX-GRT7039 compared with placebo. | Quality of life – EuroQol-5 Dimension Health Questionnaire 5<br>Levels (EQ-5D-5L): changes from baseline to Week 12,<br>Week 26, Week 38, and Week 52. |
| | Quality of life – Short form-36 (SF-36): changes from baseline to Week 12, Week 26, Week 38, and Week 52. |

# Protocol synopsis (extracted from final protocol)

Protocol KF7039-01


 DMS version 1.0 28 Oct 2021


#### Other data to be collected that are not directly attributed to an endpoint

To evaluate subject eligibility and to describe the trial population

- Demographic and other baseline characteristics: Date of signature on the informed consent form, sex, age, body weight, height, body mass index (BMI), race, ethnic group.
- Relevant prior/concomitant treatments: all prior and concomitant treatments (i.e., non-pharmacologic and pharmacologic) used to treat osteoarthritis and osteoarthritis pain and reasons for discontinuing will be collected. Prior and concomitant medications other than for osteoarthritis will be collected.
- Thorough musculoskeletal history (incl. current and past history of osteoarthritis, joint surgeries, fractures, joint injuries) and physical examination (incl. evaluation of joints for swelling, redness, tenderness).
- Imaging data (X-ray and magnetic resonance imaging [MRI]), pregnancy test, and drugs of abuse test.

#### To assess the efficacy

- Patient Global Assessment (PGA) of Osteoarthritis.
- Patient-specific functional scale (PSFS).
- WOMAC, PGIC, SF-36, and EQ-5D-5L data at time points not related to the primary and secondary endpoints.

#### To assess the safety and tolerability of RTX-GRT7039

- Vital signs (systolic and diastolic blood pressure, pulse rate, respiratory rate).
- Electrocardiogram (ECG).
- Safety laboratory parameters (hematology, clinical chemistry, clotting, and urinalysis dipstick panel).
- Physical examination findings.
- Assessment of procedural pain related to the IMP injection.
- Imaging data (X-ray and MRI).

#### To assess the treatment satisfaction

• Treatment Satisfaction Questionnaire for Medication (TSQM) scores.

### 1.3 Trial subjects – the population to be studied

Inclusion criteria are reviewed at the Screening Visit (V1) and at Baseline (i.e., V2 before IMP administration). Subjects will only receive IMP if documentation is available showing that they meet all of these inclusion criteria and none of the exclusion criteria.

#### 1.3.1 Inclusion criteria

- 1. The subject has given written informed consent to participate.
- 2. The subject is  $\ge 18$  years of age at the Screening Visit.
- 3. The subject has a BMI  $\leq 40.0 \text{ kg/m}^2$ .


Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

- 4. The subject is willing to adhere to the restricted use of concomitant treatments (see concomitant treatments in Section 1.4.3).
- 5. The subject has a diagnosis of osteoarthritis of the knee based on American College of Rheumatology criteria and functional capacity class of I to III. Pain at the index knee must be present for at least 6 months prior to Screening Visit.
- 6. The subject has a Kellgren-Lawrence (K-L) grade of 2 to 4 in the index knee (based on X-ray performed during Screening Visit, assessed by central readers).
- 7. There is a documented history indicating that subject has insufficient pain relief with optimal SoC, i.e.,
  - a. non-pharmacological treatment, and
  - b. 1 or more courses of oral non-steroidal anti-inflammatory drugs (NSAIDs) prescribed by their physician and
  - c. where appropriate opioids, intra-articular treatment with corticosteroids, and intra-articular treatment with hyaluronic acid

in combination or as monotherapies,

or subject is unable to take SoC due to contraindication or intolerability to 1 or more of the SoC treatments above.

Further details on the definition of documented history will be provided in the electronic case report form (eCRF) guidance document.

- 8. The investigator does not consider that any additional benefit can reasonably be expected from further adjustments to the subject's pain treatment.
- 9. The subject must have a baseline WOMAC pain subscale score ≥5 using the 11-point (0-10) NRS for the index knee at Screening (assessment in e-diary at V1) and at baseline (assessment in e-diary at V2).
- 10. Women of childbearing potential must have a negative pregnancy test at the Screening Visit and prior to each administration of IMP. They must also agree to practice, at a minimum, acceptable measures of birth control for at least 90 days following administration of IMP.
- 11. Male subjects agree to use barrier contraception (condom) during sexual intercourse with women of childbearing potential after each administration of IMP for 90 days. The male subject is willing to ensure that during this period the female sexual partner is additionally practicing contraception, if of childbearing potential.

#### 1.3.2 Exclusion criteria

A single re-screening is accepted for items 4, 5, 6, and 7.

- 1. The subject reports a WOMAC pain subscale score of 10 on the 11-point (0-10) NRS at Screening (assessment in e-diary at V1) or at baseline (assessment in e-diary at V2).
- 2. The subject has a WOMAC pain subscale score of ≥4 on the 11-point (0-10) NRS in the non-index knee at Screening.
- 3. The subject has past joint replacement surgery of the index knee.
- 4. The subject had an injection of either corticosteroid or intra-articular visco-supplementation (i.e., hyaluronic acid) into the index knee within 90 days of Screening.


#### Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

- 5. The subject had an injection of platelet-rich plasma or stem cells into the index knee within 6 months of Screening.
- 6. The subject applied topical capsaicin on the index knee within 3 months of Screening.
- 7. The subject has a history of significant trauma or surgery (e.g., open or arthroscopic) to the index knee within 12 months of Screening.
- 8. The subject has any known active infection, including suspicion of intra-articular infection, ulcer, or open wound anywhere on the index knee.
- 9. The subject has periarticular pain from any cause other than osteoarthritis, including referred pain, bursitis, or tendonitis.
- 10. The subject has ipsilateral clinical hip osteoarthritis on the side of the index knee.
- 11. The subject has pre-existing osteonecrosis, subchondral insufficiency fracture, atrophic osteoarthritis, severe bone on bone osteoarthritis, knee pain attributable to disease other than osteoarthritis, or the subject has rapidly progressing osteoarthritis (RPOA) Type I or Type II.
- 12. The subject has significant malalignment of anatomical axis (medial angle formed by the femur and tibia) of the target knee (varus >10, valgus >10) by X-ray as assessed by independent Central Readers at Screening Visit.
- 13. The subject has other conditions that could affect trial endpoint assessments of the index knee, including, but not limited to, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, gout or pseudogout, inflammatory bowel disease related arthropathy, peripheral neuropathy (e.g., diabetic neuropathy), lupus erythematosus, significant skin conditions overlying the index knee, acromegaly, metabolic joint diseases, and fibromyalgia.
- 14. The subject has significant pain in other areas, which may confound discrimination of pain assessment in the index knee.
- 15. The subject has evidence of cognitive impairment including dementia that may interfere with the subject's ability to complete patient reported outcomes (PROs).
- 16. The subject had systemic (except inhaled corticosteroid) immunosuppressant agent within 6 months prior to trial medication administration.
- 17. The subject has any surgery scheduled during the trial period.
- 18. The subject has current clinically significant disease(s) or condition(s) (including clinically significant cardiovascular disease) that may affect efficacy or safety assessments, or any other reason which, in the investigator's opinion, may preclude the subject's participation in the full duration of the trial.
- 19. The subject has a major bleeding disorder encompassing, but not limited to coagulopathy and any current antithrombotic and anticoagulant events.
- 20. The subject has a history of severe allergic or anaphylactic reactions.
  - The subject has a history of hypersensitivity to local anesthetic (e.g., lidocaine, ropivacaine).
  - The subject has a history of hypersensitivity to resiniferatoxin (RTX) or any similar component (capsaicin, chili peppers).
- 21. The subject has a known infection of human immunodeficiency virus, or known current acute or chronic hepatitis B or C infection.

# Protocol synopsis (extracted from final protocol)

Protocol KF7039-01

 DMS version 1.0 28 Oct 2021


- 22. The subject has unstable or poorly controlled blood pressure which, in the opinion of the investigator, would put the subject at risk of severe adverse blood pressure increases upon IMP application.
- 23. The subject has evidence or history of severe psychiatric illness/disorder during the 3 years prior to the Screening Visit that, in the investigator's opinion, may affect efficacy or safety assessments or may compromise the subject's safety during trial participation (e.g., major depression, major anxiety disorder, psychosis, severe personality disorders).
- 24. The subject has a history of alcohol or drug abuse or was actively abusing drugs (including alcohol, medication) during the 1 year prior to the Screening Visit as judged by the investigator.
- 25. The subject has past or pending litigation due to chronic pain or disability.
- 26. The subject is known or suspected of not being able to comply with the requirements of the trial protocol or the instructions of the trial site staff.
- 27. The subject is not able to communicate meaningfully with the trial site staff.
- 28. The subject is currently participating or was participating in another investigational drug trial within 3 months prior to the Screening Visit.
- 29. The subject is an employee of the investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial site or is a family member of the employees or the investigator.
- 30. The subject has contraindications to an MRI of the index knee.
- 31. The subject has a history of malignancy within 2 years prior to the Screening Visit, with the exception of basal cell carcinoma.
- 32. The female subject is pregnant, planning on becoming pregnant, or is currently breastfeeding.

#### 1.4 Trial treatments

### 1.4.1 Investigational medicinal products

The IMPs used in this trial are given below:

- 5mL RTX-GRT7039 solution for intra-articular injection is constituted from 2 vials: 1 vial containing 1.6 μg/mL RTX supplied in 0.4 mL ethanolic solution and 1 vial containing 8 mL D-α-tocopherol polyethylene glycol succinate (TPGS) buffer.
- 5 mL placebo solution for intra-articular injection is constituted from 2 vials: 1 vial containing 0.4 mL ethanolic solution (placebo to match RTX-GRT7039) and 1 vial containing 8 mL TPGS buffer.

Details will be outlined in the pharmacy manual.

A total 5 mL of IMP will be injected following ropivacaine administration (see Section 1.4.2), into the knee joint.

It is strongly recommended that the injection is assisted by ultrasound. Once completed, the needle and syringe will be removed, and an adhesive bandage applied.

The first IMP injection will occur at the Randomization Visit (V2/Day 1) and a second injection of IMP will be administered at 6 months (V6/Week 26). Re-injection is not allowed if the subject did

Grünenthal


### **Protocol synopsis** (extracted from final protocol)

Protocol KF7039-01


DMS version 1.0 28 Oct 2021

not tolerate previous IMP injection as judged by the investigator or if they developed hypersensitivity to the IMP.

#### 1.4.2 Other medication/treatments

Fifteen minutes prior to the intra-articular injection of IMP, a 5 mL intra-articular injection of ropivacaine 0.5% will be administered as a local anesthetic. Separate needles should be used for each, and the skin should be cleaned again prior to the administration of IMP.

Further details regarding the administration of ropivacaine are specified in a separate manual.

#### 1.4.3 Prohibited and allowed medications or therapies

Subjects should not receive any of the following medications or therapies for the indicated times specified below:

- Intra-articular injection of corticosteroid or intra-articular visco-supplementation (i.e., hyaluronic acid) in the index knee within 90 days before Screening and throughout the trial
- Intra-articular injection of platelet-rich plasma or stem cells into the index knee within 6 months of Screening and throughout the trial
- Topical capsaicin on the index knee within 3 months of Screening and throughout the trial
- Any surgical intervention on the index knee (including but not limited to, arthroscopic interventions and knee replacement surgery) throughout the trial
- Any other investigational treatment or therapy

Subjects should continue their baseline non-pharmacological treatments and baseline analgesic and osteoarthritis medication(s) as long as the medications are not prohibited as outlined below, if they are on a stable, well-defined treatment regimen for at least 1 month before allocation to IMP and are anticipated to be able to maintain the treatment regimen in the opinion of the investigator.

There should be no changes (increases, decreases, or switches) from or additions to baseline analgesic medications (NSAIDs, opioids, other) and nonpharmacologic treatments after the Screening Visit. This is designed to minimize possible confounding treatment effects due to alterations in pain medications.

Furthermore, subjects should not schedule any medical procedures which would likely require an adjustment in pain medications during the trial and in particular for Weeks 10 to 12, Weeks 24 to 26, Weeks 36 to 38, and Weeks 50 to 52, if possible. Subjects not taking opioids at baseline should similarly refrain from starting opioid treatment.

If for any reason deemed necessary by the investigator, a subject requires additional medication(s) or change of dose, the medication(s), dosage change, route of administration, start and stop dates, and the indication for which it was given must be recorded in the source documents and a specific page in the eCRF.

All vaccinations, including Coronavirus disease 2019 (COVID-19), are permitted during the trial.

#### 1.5 Statistical analyses

All statistical methods will be detailed in a statistical analysis plan (SAP). The SAP will be finalized prior to database lock and unblinding.

Grünenthal


# Protocol synopsis (extracted from final protocol)

Protocol KF7039-01


 DMS version 1.0 28 Oct 2021

## 1.5.1 Sample size rationale

Effect size estimates were based on relevant literature and the results of available MTX-071-P03 trial results utilizing the absolute change from baseline to Week 12 endpoint. A total number of 382 subjects are required to achieve an overall power of at least 90% to reject the null hypothesis of no treatment difference in treatment group means between RTX-GRT7039 and placebo (2-sided t-test, type I error of  $\alpha = 0.05$ ). This is based upon an expected treatment difference of at least 1 point on 11-point (0-10) NRS (absolute change from baseline in the WOMAC pain subscale score) on the primary efficacy endpoint and a standard deviation of 3 in both treatment groups.

To be able to conduct confirmatory testing for the secondary endpoints, an alpha-adjustment will need to be taken into consideration. The sample size is, therefore, expected to be approximately a total of 450 subjects (225 on placebo and 225 on RTX-GRT7039) including no more than 90 subjects from Japan.

Assuming a screening failure rate of about 40%, approximately 750 subjects are planned to be screened to randomize 450 subjects for the primary analysis (225 evaluable subjects for the RTX-GRT7039 treatment arm, and 225 for the placebo arm, 1:1 randomization).

### 1.5.2 Subject populations

#### Safety Analysis Set

Defined as all subjects with at least 1 IMP administration (including incomplete administrations).

Analyses on the Safety Analysis Set (SAF) will be conducted based on actual treatment received.

### **Full Analysis Set**

Defined as all randomly assigned subjects with at least 1 IMP administration (including incomplete administrations).

Analyses on the Full Analysis Set (FAS) will be conducted based on the treatment as randomized (i.e., based on planned treatment).

### 1.5.3 Statistical methods and analysis

To evaluate the primary endpoint, the WOMAC pain subscale with a 48-hour recall period will be assessed weekly using e-diaries. The WOMAC pain subscale is comprised of 5 questions regarding the amount of pain experienced due to osteoarthritis in the index knee in the past 48 hours using an 11-point (0-10) NRS. The WOMAC pain subscale score will be calculated as the mean of the non-missing scores from the 5 individual questions, which may not be a whole (integer) number. The baseline WOMAC pain subscale score is defined as the assessment made at the Randomization Visit (V2).

The estimand of interest for the primary efficacy analysis is the difference in mean change from baseline in 48-hour WOMAC pain subscale score at Week 12 in the index knee using an 11-point (0-10) NRS between RTX-GRT7039 and placebo, in subjects who initiate treatment, as if substantial changes in background medication or addition of new analgesics were not available.

The primary efficacy analysis will be performed using a mixed-effects model for repeated measures (MMRM). The model will include fixed effects of treatment, country/region, gender, time (corresponding to trial week), and treatment-by-time interaction. The baseline value will be a

DMS version: 1.0

ID: 1423148

Protocol synopsis 

## (extracted from final protocol)

Grünenthal

Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

covariate. Time will be included in the MMRM analysis to account for the correlation in repeated measures within-subject. An unstructured [UN] covariance matrix will initially be fitted to the MMRM. In the event that the analysis model does not converge, then the Toeplitz (TOEP) will be used as the covariance matrix. The auto-regressive (1) [AR(1)] covariance matrix will be used if TOEP also fails to converge. In the event that AR(1) also results in non-convergence, the compound symmetry covariance matrix [CS] will be used.

Individual sites will be pooled by geographic region. Geographic regions will be defined in the SAP and correspond to the country/region used in the stratified randomization.

For the primary analysis the following intercurrent events (IE) will be considered:

- A substantial change in the analgesic osteoarthritis background therapy (optimal SoC) will be considered as an IE. For this, a hypothetical policy estimand strategy is applied. Values after the occurrence of the IE will be excluded from the analyses and will be imputed by the baseline value.
- Any other substantial change in analgesic medication given for any other indication will be considered an IE. For this, a hypothetical policy estimand strategy is applied. Values after the occurrence of the event will be excluded from the analyses and will be imputed by the last observation.
- For the analyses on Week 52 endpoints, not having received a second dose of treatment is considered an IE. For this, a hypothetical policy estimand strategy is applied. Values after the occurrence of the IE will be imputed by the last observation or, at the latest, the Week 26 value.

Sensitivity analyses will be performed.

Subgroup analyses may be considered if appropriate and will be specified in the SAP.

#### 1.5.4 Interim analysis

No interim analyses are planned for this trial.


Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

## 1.6 Schedule of events

| Trial Period | Screening Period | Treatment and Follow-up Period | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1<br>(Screening Visit) | V2 <sup>a</sup><br>(Randomization<br>Visit) | V3<br>± 3<br>days | V4<br>± 3<br>days | V5<br>±7<br>days | V6 <sup>a</sup><br>± 3 days | V7<br>± 3<br>days | V8<br>± 3<br>days | V9<br>±7 days | V10<br>Final Visit/Early<br>Termination Visit <sup>b</sup><br>± 7 days |
| Day | -30 to -1 | 1 | 8 | 29 | 85 | 183 | 190 | 211 | 267 | 365 |
| Week | | | 1 | 4 | 12 | 26 | 27 | 30 | 38 | 52 |
| Obtain informed consent | X | | | | | | | | | |
| Collect demographic data | X | | | | | | | | | |
| Record general and musculoskeletal specific medical history <sup>c</sup> | X | | | | | | | | | |
| Record prior medications/therapies <sup>c</sup> | X | | | | | | | | | |
| Record concomitant medications/therapies | X | X | X | X | X | X | X | X | X | X |
| Perform physical exam | X | X | X d | X d | X d | X | X d | X d | X d | X |
| Record vital signs | X | X | X e | X e | X | X | X e | X e | X | X |
| Perform scheduled X-rays of index knee | X f | | | | | X | | | | X |
| Perform MRI of the index knee <sup>g</sup> | X h | | | | | | | | | |
| ECG | X | X | | | | X | | | | X |
| Check inclusion/exclusion criteria | X | X | | | | | | | | |
| Train subjects on e-diaries | X | | | | | | | | | |

### 

# Protocol synopsis (extracted from final protocol)

### Grünenthal


Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

| Trial Period | Screening Period | eening Period Treatment and Follow-up Period | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1<br>(Screening Visit) | V2 <sup>a</sup><br>(Randomization<br>Visit) | V3<br>± 3<br>days | V4<br>± 3<br>days | V5<br>±7<br>days | V6 <sup>a</sup><br>± 3 days | V7<br>± 3<br>days | V8<br>± 3<br>days | V9<br>±7 days | V10<br>Final Visit/Early<br>Termination Visit <sup>b</sup><br>± 7 days |
| Day | -30 to -1 | 1 | 8 | 29 | 85 | 183 | 190 | 211 | 267 | 365 |
| Week | | | 1 | 4 | 12 | 26 | 27 | 30 | 38 | 52 |
| Dispense e-diary | X | | | | | | | | | |
| Placebo response reduction training and accurate pain reporting training for subjects | X | | | | X | X | | | X | |
| Ask subject to record WOMAC pain subscale score in the non-index knee in their e-diary | X | | | | | | | | | |
| Ask subject to record WOMAC assessments for the index knee in their e-diary i | X | X | X | X | X | X | X | X | X | X |
| Check e-diary compliance j | X | X | X | X | X | X | X | X | X | X |
| Dispense subject trial card | X | | | | | | | | | |
| PGIC | | | | | X | X | | | X | X |
| PGA | | X | X | X | X | X | X | X | X | X |
| PSFS | | X | X | X | X | X | X | X | X | X |
| EQ-5D-5L | | X | X | X | X | X | X | X | X | X |
| SF-36 | | X | | | X | X | | | X | X |
| TSQM | | | | | X | X | | | X | X |

#### 

# Protocol synopsis (extracted from final protocol)

### Grünenthal


Protocol KF7039-01

 DMS version 1.0 28 Oct 2021

| Trial Period | Screening Period | Treatment and Follow-up Period | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1<br>(Screening Visit) | V2 <sup>a</sup><br>(Randomization<br>Visit) | V3<br>± 3<br>days | V4<br>± 3<br>days | V5<br>±7<br>days | V6 <sup>a</sup><br>± 3 days | V7<br>± 3<br>days | V8<br>± 3<br>days | V9<br>±7 days | V10<br>Final Visit/Early<br>Termination Visit <sup>b</sup><br>± 7 days |
| Day | -30 to -1 | 1 | 8 | 29 | 85 | 183 | 190 | 211 | 267 | 365 |
| Week | | | 1 | 4 | 12 | 26 | 27 | 30 | 38 | 52 |
| Collect urine and perform pregnancy (if applicable) and drugs of abuse testing | X | X | | | | $X^k$ | | | | |
| Safety laboratory | X | X | | | | X | | | | X |
| Randomization to treatment | | X | | | | | | | | |
| Pre-treatment with ropivacaine intra-articular injection | | X | | | | X | | | | |
| Intra-articular IMP injection | | X | | | | X | | | | |
| Ask subjects to rate their procedural pain <sup>1</sup> | | X | | | | X | | | | |
| Record adverse events m | X | X | X | X | X | X | X | X | X | X |
| Collect e-diary | | | | | | | | | | X |
| Collect subject trial card | | | | | | | | | | X |

- a) All other assessments are completed prior to IMP administration, assessment of procedural pain, and recording of adverse events.
- b) Subjects who discontinue or are discontinued earlier from the trial will perform the Final Visit/Early Termination Visit as a last trial visit, if possible.
- c) At Screening, a comprehensive musculoskeletal medical history is obtained. History of insufficient pain relief, inability to tolerate or contraindication to take the specified SoC treatments should be collected. Any prior use of medication used to treat osteoarthritis and osteoarthritis pain and prior use for all other medications should be collected.
- d) Physical examination of only the index knee at specified visits.
- e) Body weight and BMI are not recorded at these visits

# Protocol synopsis (extracted from final protocol)

Grünenthal


Protocol KF7039-01


 DMS version 1.0 28 Oct 2021

- f) To be performed at V1 or between V1 and V2, only if all inclusion criteria and no exclusion criteria that can be evaluated at Screening are met.
- g) Follow up MRIs may be performed in case of index knee related adverse events or unexpected increased pain scores of severe intensity, which are persistent for at least 2 weeks despite treatment with analgesic medication according to investigator judgment.
- h) At V1 or between V1 and V2, only if all inclusion criteria and no exclusion criteria that can be evaluated at Screening are met. Use of historical MRI 30 days before Screening is acceptable, if no relevant change in pain occurred since then (according to investigator and subject judgement).
- i) In the first week after an intra-articular IMP injection (i.e., Day 1 to 7 and Week 26), subjects will assess the WOMAC pain and physical function subscales with 48-hour recall period every 2 days. After the first week post IMP injection, the WOMAC pain subscale score will continue to be assessed weekly in the e-diary and the complete WOMAC will be assessed and recorded in the subject's e-diary at the visits specified in this SoE.
- j) Starting after V1, until V10 the e-diary will be reviewed for completeness prior to initiating any treatment-associated procedures. The subject will be re-trained if needed.
- k) Urine pregnancy test only at this visit, if applicable.
- 1) Subjects will be asked to rate their procedural pain (current pain intensity on the 11-point [0-10] NRS) using the tablet computer at the site at the following time points: -0.5, 0, 0.5, 1, 1.5, and 3 hours relative to intra-articular IMP injections, with time point 0 immediately before IMP injection.
- m) Adverse events of sensory loss and decrease of motor function at the index knee/the leg of the index knee should be evaluated by additional physical examinations, X-rays, MRIs as deemed required by the investigator.

BMI = body mass index; ECG = electrocardiogram; e-diary = electronic diary; EQ-5D-5L = EuroQol-5 Dimension Health Questionnaire 5 Levels; exam = examination; IMP = investigational medicinal product; MRI = magnetic resonance imaging; NRS=numeric rating scale; PGIC = Patient Global Impression of Change; PGA = Patient Global Assessment of Osteoarthritis; PSFS = Patient Specific Functional Scale; SF-36 = Short Form-36 Health Survey; SoC = standard of care; SoE = schedule of events; TSQM = Treatment Satisfaction Questionnaire for Medication; V = Visit; WOMAC = Western Ontario and McMaster Universities Osteoarthritis Index.